CLINICAL TRIAL: NCT01995877
Title: Evaluation of the Influence of Body Position on the Inferior Vena Cava (IVC) Diameter
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment, PI leaving university
Sponsor: University of Michigan (Other)
Collaborators: Bard Ltd (Industry)
Responsible Party: Principal Investigator, Ranjith Vellody, Principal Investigator, University of Michigan
Other Study IDs: HUM00034464
Record Dates: First submitted 2013-11-21; First posted 2013-11-27 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Vena Cava Filters

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subjects scheduled for IVC filter placement: A filter may be needed to be placed in the IVC (inferior vena cava) to prevent blood clots from traveling from legs to lungs. Patients who have had a pelvic fracture, or have blood clots in the leg(s) may need an IVC. Filter placement may be ordered when a patient is scheduled for major surgery and extensive bed rest.
  Interventions: Procedure: Subjects scheduled for IVC filter placement

INTERVENTIONS:
Procedure: Subjects scheduled for IVC filter placement — Subjects will have an intra vascular ultrasound (IVUS) performed while lying down on the exam table; this will be performed before and after the IVC (inferior vena cava) filter is placed. During the ultrasound, measurements of the diameter of different areas of the IVC will be taken. The table will then be moved so that you are in a standing position and the measurements will be taken again.
  The ultrasound will be done by the physician performing your procedure. When you are lying down, a sheath (small catheter) will be inserted into a vein in your groin. The IVUS (intra vascular ultrasound) catheter will be inserted through the sheath and used to measure the size of the IVC at various places.
  The IVUS procedure will add about 30-45 minutes to the filter placement procedure.
  Other Names: IVUS(intra vascular ultrasound)

SUMMARY:
To determine if laying down or standing up changes the diameter of the inferior vena cava.

DETAILED DESCRIPTION:
Patients are referred for IVC(inferior vena cava)filter placement secondary to trauma, surgery, a fractured pelvis or known blood clots in the lower extremities. The filter is placed to prevent blood clots from traveling into the lungs. The filters are placed during a interventional radiology procedure. During the procedure the diameter of the IVC(inferior vena cava)is measured with the patient in a horizontal position (laying down). The blood pressure in the IVC when a patient is in this position is relatively low in normal circumstances, but may increase substantially when the patient is vertical with secondary dilation of the IVC(inferior vena cava).

Migration of IVC(inferior vena cava)filters is not frequent; however it is a serious complication, which may be caused by changes in the diameter of the IVC(inferior vena cava)related to changes in the position of the body and/or increased pressure in the abdomen.

The purpose of this study is to evaluate how much postural changes of the body affect the diameter of the IVC(inferior vena cava).

For research purposes patients will have an intravascular ultrasound (IVUS) performed to measure the IVC diameter before and after a Valsalva maneuver (having the subject hold their breath and bear down as if they were having a bowel movement). The angiographic table will be elevated and the measurements will be repeated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. Subjects who will have a clinically indicated IVC filter placement procedure scheduled.
3. Only subjects with no contraindications to being elevated up to a standing or near standing position on the angiography table.

   -

Exclusion Criteria:

1. Pregnant
2. Have a broken leg or any other physical condition that won't allow you to stand.
3. If you are in a traction device
4. If you have a brain injury and require special monitoring of the pressure in the brain.
5. Patients on a ventilator cannot participate in this study.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are receiving an IVC(inferior vena cava) filter as part of their standard therapy.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Body postural changes and the effect on the diameter of the inferior vena cava. | 45 minutes
  Migration of IVC filters is not frequent; however it is a serious complication, which may be caused by changes in the diameter of the IVC related to changes in the position of the body and/or increased pressure in the abdomen.
  The purpose of this study is to evaluate how much postural changes of the body affect the diameter of the IVC.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjith Vellody, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No